CLINICAL TRIAL: NCT07088354
Title: Deep Learning Model Predicts Pathological Complete Response of Esophageal Squamous Cell Carcinoma Following Neoadjuvant Immunochemotherapy
Acronym: DL-ESCC
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Yangkai Li, professor, Tongji Hospital
Other Study IDs: ESRA-01
Record Dates: First submitted 2025-07-17; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Immunochemotherapy; Pathological Complete Response; Deep Learning
Keywords: Esophageal Squamous Cell Carcinoma; Neoadjuvant Immunochemotherapy; Deep Learning; Pathological Complete Response
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- ESCC Patients Undergoing Neoadjuvant Immunochemotherapy and Surgery: Patients with esophageal squamous cell carcinoma treated with neoadjuvant immunochemotherapy followed by surgery.
  Interventions: Diagnostic Test: The high-throughput extraction of large amounts of quantitative image features from medical images

INTERVENTIONS:
Diagnostic Test: The high-throughput extraction of large amounts of quantitative image features from medical images — The high-throughput extraction of large amounts of quantitative image features from medical images

SUMMARY:
This study aims to develop and validate a deep learning model to predict pathological complete response (pCR) in patients with esophageal squamous cell carcinoma who have undergone neoadjuvant immunochemotherapy. Clinical, imaging, and pathological data from previously treated patients will be collected and analyzed. The model is expected to assist in predicting treatment outcomes and guide personalized therapeutic strategies.

DETAILED DESCRIPTION:
This multicenter retrospective study will collect chest CT images and clinical data from patients with esophageal squamous cell carcinoma (ESCC) who underwent surgery following neoadjuvant immunochemotherapy between January 2019 and July 2025. Deep learning features will be extracted from the CT images to develop a predictive model of pathological complete response (pCR). The model's performance will be evaluated using metrics including the area under the receiver operating characteristic curve (AUC), accuracy, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV). Additionally, SHapley Additive exPlanations (SHAP) analysis will be employed to quantify the contribution of CT imaging features to the model's predictions. This study aims to improve early identification of responders to neoadjuvant immunochemotherapy and support personalized treatment strategies for ESCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed esophageal squamous cell carcinoma (ESCC).
2. Received at least one cycle of neoadjuvant chemotherapy combined with immunotherapy.
3. Underwent contrast-enhanced chest CT before initiation of neoadjuvant treatment.
4. Underwent contrast-enhanced chest CT after completion of neoadjuvant treatment and prior to surgery.

Exclusion Criteria:

1. Diagnosis of other malignancies.
2. Received other anti-tumor therapies before or during neoadjuvant chemo-immunotherapy.
3. Incomplete clinical data.
4. Poor-quality CT imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with esophageal squamous cell carcinoma who received at least one cycle of neoadjuvant chemotherapy combined with immunotherapy, with available contrast-enhanced chest CT scans before and after neoadjuvant treatment, and who underwent surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | Assessed at the time of surgery, within 1 month post-treatment.
  The proportion of patients achieving complete pathological remission after neoadjuvant immunochemotherapy followed by surgery.

SECONDARY OUTCOMES:
Model Performance Metrics (AUC, Accuracy, Sensitivity, Specificity, PPV, NPV) | At the time of model validation, approximately one year on average after the completion of the research.
  Evaluation of the deep learning model's predictive performance using receiver operating characteristic curve (AUC), accuracy, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Overall Officials: Yangkai Li, MD, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No